CLINICAL TRIAL: NCT01908894
Title: A Double-blind Study of the Pharmacokinetic and Pharmacodynamic Properties of BIOD-123 and BIOD-125 Compared to Humalog® in Subjects With Type 1 Diabetes Including Assessments of Safety and Injection Site Toleration
Brief Title: Pharmacokinetic and Pharmacodynamic Properties of BIOD-123 and BIOD-125 Compared to Humalog® in Subjects With Type 1 Diabetes Including Assessments of Injection Site Toleration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biodel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 3-101
Record Dates: First submitted 2013-07-24; First posted 2013-07-26 (Estimated); Last update posted 2013-07-26 (Estimated); Status verified 2013-07

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Insulin Lispro

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- BIOD-123 (Experimental): SC administration of 0.20 U/kg
  Interventions: Drug: BIOD-123
- BIOD-125 (Experimental): SC administration of 0.20 U/kg
  Interventions: Drug: BIOD-125
- Humalog (Active Comparator): SC administration of 0.20 U/kg
  Interventions: Drug: Humalog

INTERVENTIONS:
Drug: BIOD-123
  Arms: BIOD-123
Drug: BIOD-125
  Arms: BIOD-125
Drug: Humalog
  Arms: Humalog

SUMMARY:
The primary objective is to assess the speed of absorption of BIOD-123 and BIOD-125 and compare them to Humalog.

DETAILED DESCRIPTION:
The primary objective is to assess the speed of absorption of BIOD-123 and BIOD-125 and compare them to Humalog.

The secondary objectives are to assess other pharmacokinetic characteristics of BIOD-123 and BIOD-125 and compare those to Humalog®, to assess pharmacodynamic characteristics of BIOD-123 and BIOD-125 and compare those to Humalog®, and to evaluate the safety and tolerability of BIOD-123 and BIOD-125 compared to Humalog®

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥18 - ≤70 years
2. BMI: ≥18 - ≤30 kg/m2
3. Diagnosed with type 1 diabetes mellitus for at least 1 year
4. Insulin antibody ≤10 μU/mL at screening

Exclusion Criteria:

1. Type 2 diabetes mellitus
2. History of >2 severe hypoglycemic events within the 3 months prior to screening
3. Serum C-peptide >1.0 ng/mL
4. Hemoglobin A1c (HbA1c) >10.0%
5. Females who were breast feeding, pregnant, or intending to become pregnant during the study
6. A sexually active person who was not using adequate contraceptive methods
7. Positive serology for human immunodeficiency virus (HIV), Hepatitis B, or Hepatitis C
8. Abnormal ECG, safety lab, or physical examination results that were deemed clinically significant by the investigator

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-02; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Speed of absorption (TINS-50%-early) of BIOD-123 and BIOD-125 versus Humalog. | 0-30, 0-60, 0-90, 0-480, and 120-480 minutes
  Subjects were to receive study drug at 3 separate dosing visits separated by 3-28 days. The estimated duration of study participation for 1 subject was approximately 12 weeks. The estimated duration of the study was approximately 6 months.